CLINICAL TRIAL: NCT02991248
Title: Improve Dynamic Lateral Balance of Humans With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Ming Wu, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD083314 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-12-13 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- robotic training & stimulation (Experimental): Device: robotic treadmill training paired with active spinal cord electrical stimulation, three times a week for 6 weeks.
  Interventions: Device: robotic training; Device: spinal cord electrical stimulation; Device: treadmill
- robotic training & sham (Active Comparator): Device: robotic training paired with sham spinal cord stimulation, three time a week for 6 weeks.
  Interventions: Device: robotic training; Device: treadmill
- treadmill only (Placebo Comparator): Device: treadmill Conventional treadmill training only, three time a week for 6 weeks.
  Interventions: Device: treadmill

INTERVENTIONS:
Device: robotic training — robotic training by applying pelvis force perturbation
  Arms: robotic training & sham; robotic training & stimulation
Device: spinal cord electrical stimulation — Applying direct current electrical stimulation on spinal cord
  Arms: robotic training & stimulation
Device: treadmill — conventional treadmill training only

SUMMARY:
This study is to test whether pelvis perturbation training paired with transcutaneous spinal direct current stimulation (tsDCS) will be effective in improving dynamic balance and locomotor function in humans with SCI. One group will receive pelvis perturbation training paired with tsDCS, one group will receive pelvis perturbation training paired with sham, and one group will receive treadmill training only.

DETAILED DESCRIPTION:
A major goal of patients with spinal cord injury (SCI) is to regain walking ability, as limitations in mobility can affect most activities of daily living. In addition, patients with SCI may experience a higher incidence of falls due to impaired balance and gait. Dynamic balance control plays a crucial role during locomotion in human SCI. Thus, improved dynamic balance may facilitate locomotion in this population. Current balance training paradigms can be effective in improving balance during standing, but are less effective in improving dynamic balance during locomotion in humans with SCI. Thus, there is a need to develop new paradigms for improving dynamic balance and locomotor function in patients with SCI. The goal of this study is to test whether pelvis perturbation training paired with transcutaneous spinal direct current stimulation (tsDCS) will be effective in improving dynamic balance and locomotor function in humans with SCI. We postulate that providing a perturbation force to the pelvis during treadmill training will increase the activation of muscles used for maintaining lateral balance while walking. Further, repeated activation of particular sensorimotor pathways may reinforce circuits and synapses used for lateral balance control through a use-dependent neural plasticity mechanism. However, the excitability of spinal cord neural circuitries may be depressed due to the reduced descending drive signals from the upper level control center after SCI, which may reduce the efficacy of neuralplastic changes achieved following rehabilitation. The excitability of neural pathways is crucial for neural reorganization achieved following rehabilitation. Recently studies indicate that tsDCS may modulate the excitability of neural circuitries of the spinal cord in patients with SCI. Thus, we postulate that controlled pelvis perturbation training paired with tsDCS will be more effective than that paired with a sham in improving dynamic balance and locomotor function in humans with SCI. Results obtained from this study will lead to an innovative clinical therapy aimed at improving balance and walking function in humans with SCI. Improvements in balance and walking function may allow for increased participation in community-based ambulation and activities, and significantly improve quality of life in humans with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;
2. medically stable with medical clearance to participate;
3. level of the SCI lesion between C4-T10;
4. passive range of motion of the legs within functional limits of ambulation;
5. ability to walk on a treadmill for more than 20 minutes with partial body weight support as needed and short sitting/standing breaks;
6. ability to ambulate without orthotics or with orthotics that do not cross the knee for more than 10 meters

Exclusion Criteria:

1. the presence of unhealed decubiti, existing infection, severe cardiovascular and pulmonary disease, concomitant central or peripheral neurological injury (e.g. traumatic head injury or peripheral nerve damage in lower limbs);
2. history of recurrent fractures and/or known orthopedic injury to the lower extremities;
3. Botox injection within 6 months of starting the study, and current receiving physical therapy treatment;
4. have metallic implantation in the spinal region underneath where electrodes may be placed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in overground gait speed from baseline | post 6 weeks of training and 8 weeks after the end of training
  gait speed

SECONDARY OUTCOMES:
Changes in balance (BBS score) from baseline | post 6 weeks of training and 8 weeks after the end of training
  Berg Balance Score
Changes in dynamic gait index from baseline | post 6 weeks of training and 8 weeks after the end of training
  Dynamic Gait Index
Changes in 6 minutes walking distance from baseline | post 6 weeks of training and 8 weeks after the end of training
  Walking distance in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wu, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Abilitylab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes